CLINICAL TRIAL: NCT06296173
Title: Open Lung Protective Extubation Following General Anesthesia: the OLEXT-3 Trial
Brief Title: Open Lung Protective Extubation Following General Anesthesia
Acronym: OLEXT-3
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Collaborators: CHU de Quebec-Universite Laval (Other); The Ottawa Hospital (Other); University Health Network, Toronto (Other); Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MP-02-2024-12094
Record Dates: First submitted 2024-02-21; First posted 2024-03-06 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2025-01

CONDITIONS: Intra-abdominal Surgery; Anesthesia; Lung Injury; Ventilator-Induced Lung Injury; Atelectasis
MeSH Terms: conditions — Lung Injury; Ventilator-Induced Lung Injury; Pulmonary Atelectasis

STUDY DESIGN:
Intervention Model Description: During surgical closure, the definitive ARISCAT score and exclusion criteria will be assessed. Patients will be randomized equally (1:1) using web-based allocation-concealed methods, with stratification by center and ARISCAT risk category. An unblinded research assistant will reveal group allocation to the anesthesiologist and monitor the emergence procedure.
Who Masked: Participant, Outcomes Assessor
Masking Description: Until surgical closure, all will be blinded to treatment allocation. Only specific healthcare professionals (anesthesiologist, respiratory therapist, operating room nurses, unblinded research assistant) will be present during emergence to maintain blinding. Other healthcare team members will remain blinded. Outcome adjudicators, Executive and Steering committee members, and the data analyst will also be blinded. No mechanism for unblinding is planned, as both interventions follow the same diagnostic and treatment algorithms for adverse effects.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Open lung extubation (Experimental): At the beginning of emergence, patients will be positioned with the head of the bed elevated to at least 30 degrees and the FiO2 will be set at 50%. At the resumption of spontaneous ventilation or earlier at the discretion of the anesthesiologist, the ventilator will be set to pressure support ventilation mode for the rest of the emergence procedure. The pressure support level will be adjusted to obtain a volume similar to the one used prior to emergence. PEEP will be left unchanged. Anesthesiologists will be instructed not to switch off the ventilator until the patient is extubated.
  Interventions: Other: Protective "open-lung" extubation
- Conventional extubation (Active Comparator): At the beginning of emergence, patients will be positioned in a dorsal decubitus position and the FiO2 will be set at 100%. At the resumption of spontaneous ventilation or earlier at the discretion of the anesthesiologist, the ventilator will be switched off for the rest of the emergence procedure with the adjustable pressure-limiting valve open to atmosphere. Manual ventilation or assistance will be allowed, but the adjustable pressure-limiting valve will be reopened when pausing manual ventilation or assistance.
  Interventions: Other: Conventional extubation

INTERVENTIONS:
Other: Protective "open-lung" extubation — Emergence using 50% FiO2, semi-sitting position with pressure support ventilation and preserved PEEP
  Arms: Open lung extubation
Other: Conventional extubation — Emergence using 100% FiO2, dorsal decubitus position with assistance or manual bag ventilation without PEEP
  Arms: Conventional extubation

SUMMARY:
Perioperative respiratory complications are a major source of morbidity and mortality. Postoperative atelectasis plays a central role in their development. Protective "open lung" mechanical ventilation aims to minimize the occurrence of atelectasis during the perioperative period. Randomized controlled studies have been performed comparing various "open lung" ventilation protocols, but these studies report varying and conflicting effects. The interpretation of these studies is complicated by the absence of imagery supporting the pulmonary impact associated with the use of different ventilation strategies. Imaging studies suggest that the gain in pulmonary gas content in "open lung" ventilation regimens disappears within minutes after the extubation. Thus, the potential benefits of open-lung ventilation appear to be lost if, at the time of extubation, no measures are used to keep the lungs well aerated. Recent expert recommendations on good mechanical ventilation practices in the operating room conclude that there is actually no quality study on extubation.

Extubation is a very common practice for anesthesiologists as part of their daily clinical practice. It is therefore imperative to generate evidence on good clinical practice during anesthetic emergence in order to potentially identify an effective extubation strategy to reduce postoperative pulmonary complications.

DETAILED DESCRIPTION:
The aim of this study is to establish the feasibility of a multicenter randomized controlled clinical trial comparing two clinical strategies called "open lung" and "conventional" during extubation. The investigators also aim to estimate the rates of postoperative pulmonary complications in the two intervention groups.

METHODS

A multicenter internal pilot, prospective, randomized, allocation-concealed and controlled assessor-blinded study. Two hundred sixteen patients scheduled to undergo elective intra-abdominal surgery requiring general anesthesia and planned hospitalization at four Canadian hospitals, and at moderate or high risk of postoperative pulmonary complications according to the ARISCAT score will be recruited. Following the administration of standardized mechanical ventilation and after obtaining consent, participants will be randomly assigned to two groups:

Group A: Intervention group, "open lung" extubation strategy Group B: Control group, "conventional" extubation strategy.

The rate of adherence to the extubation protocol, the weekly patient recrutement rate and the 7-day postoperative pulmonary complications outcome completion rate will be measured. We will only report secondary efficacy outcome in aggregate as they will be rolled over to the definitive trial.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (18 years of age or over)
* Elective intra-abdominal surgery under general anesthesia.
* Moderate or high risk of postoperative pulmonary complication according to the ARISCAT score (score of 26 or more)
* Planned postoperative hospitalization

Exclusion Criteria:

* Expected or known difficult intubation according to the treating anesthesiologist
* Postoperative mechanical ventilation (planned or unplanned)
* General anesthesia performed outside the main operating room

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 270 (Estimated)
Dates: Start 2024-10-08 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2027-04-01 (Estimated)

PRIMARY OUTCOMES:
Average weekly patient recruitment rate | Every week. At the end of the study (average 9 months) at the study level.
  Achieve a weekly patient recruitment rate of 2 patients per week per center
Protocol adherence rate | At the end of surgery for individual assessments. At the end of the study (average 9 months) at the study level.
  Assess adherence to a protocol during emergence from anesthesia, monitoring four criteria (proper positioning (dorsal decubitus or semi-sitting position), correct FiO2 (100% or 50%), appropriate ventilatory mode (manual or pressure support ventilation), and proper end-expiratory pressure (zero or preserved end-expiratory pressure), and noting deviations, with adherence defined as successful performance of all criteria during extubation.
Postoperative pulmonary complications outcome completion rate | At postoperative day 7 for individual assessments. At the end of the study (average 9 months) at the study level.
  Postoperative pulmonary complications are defined as a composite endpoint that includes atelectasis, pneumonia, acute respiratory distress syndrome, and pulmonary aspiration, according to the StEP-COMPAC definition.

SECONDARY OUTCOMES:
Accuracy of self-reported protocol adherence compared to directly observed protocol adherence | At the end of the surgery
  Following emergence from general anesthesia, treating anesthesiologists will complete the same four-point scoring sheet as the research assistant to self-report protocol adherence.
Postoperative pulmonary complications | At postoperative day 7
  Postoperative pulmonary complications are defined as a composite endpoint that includes atelectasis, pneumonia, acute respiratory distress syndrome, and pulmonary aspiration, according to the StEP-COMPAC definition.
Amount of supplemental oxygen administered following discharge from the post-anesthesia care unit | At postoperative day 7 or hospital discharge (earliest of the two)
  Obtained from the electronic medical record or the handwritten vital signs sheet. Calculated as %.h-1
Quality of recovery | At postoperative day 1
  Evaluated using the QoR-15 questionnaire completed at the bedside.
Discharge disposition | At postoperative day 30
  Location to which patient is discharged (e.g., home, long term care facility, etc.) Assessed during telephone interview and using administrative data. We will
Days alive and out of hospital | At postoperative day 30
  Assessed during telephone interview and using administrative data
Health-related quality of life | At postoperative day 90
  Evaluated using the EQ-5D-5L questionnaire completed during a telephone interview

OTHER OUTCOMES:
Lowest oxygen saturation post-extubation in the operating room | At operating room exit
  Lowest SpO2 in the operating room during emergence
Time in minutes with oxygen saturation < 85% post-extubation in the operating room | At operating room exit
  Time with SpO2 < 85% in the operating room during emergence
Re-intubation rate in the operating room and in the post-anesthesia care unit | At discharge from the post-anesthesia care unit
  Re-intubation in the operating room during emergence or in the post-anesthesia care unit

CONTACTS AND LOCATIONS:
Overall Officials: Martin Girard, MD, Principal Investigator — Centre hospitalier de l'Université de Montréal (CHUM)
Locations (4):
- Canada (4):
  - The Ottawa Hospital, Ottawa, Ontario
  - Unity Health Network, Toronto, Ontario
  - Centre Hospitalier de l'Université de Montréal (CHUM), Montreal, Quebec
  - CHU de Québec - Université Laval, Québec, Quebec

IPD SHARING:
Plan to Share IPD: No
End-of-grant knowledge translation modalities will be used to reach other important stakeholders, researchers and members of the anesthesia community: scientific meetings, open access publication in a Canadian journal, and public presentations with patient partners. Knowledge diffusion on potential difficulties of conducting such trials (and solutions) will be transferred to the research community through meetings of the Canadian Perioperative Anesthesia Clinical Trial group (PACT). A methodological meeting will be organized with participating sites of both pilot and future efficacy phases to enhance protocol applicability before going forward to the efficacy phase. This plan will help recruit more Canadian centres for the efficacy trial and conduct the intervention in these centres.